CLINICAL TRIAL: NCT01509846
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Immunogenicity of an Oral Inactivated Whole Cell Shigella Flexneri 2a Vaccine in Healthy Adult Subjects
Brief Title: Safety Study of Inactivated Shigella Whole Cell Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAC 001
Record Dates: First submitted 2012-01-05; First posted 2012-01-13 (Estimated); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Shigellosis
Keywords: Shigella; vaccine; shigellosis; dysentery; whole cell
MeSH Terms: conditions — Dysentery, Bacillary; Dysentery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): Received one oral dose of 2.6±0.8 x 10^8 vp/mL Shigella flexneri 2a whole cell killed vaccine (Sf2aWC)
  Interventions: Biological: Vaccine: 2.6±0.8 x 10^8 vp/mL, 1 dose
- Cohort 2 (Experimental): Received three oral doses of 2.6±0.8 x 10^9 vp/mL Shigella flexneri 2a whole cell killed vaccine (Sf2aWC)
  Interventions: Biological: Vaccine: 2.6±0.8 x 10^9 vp/mL, 3 doses
- Cohort 3 (Experimental): Received three oral doses of 2.6±0.8 x 10^10 vp/mL Shigella flexneri 2a whole cell killed vaccine (Sf2aWC)
  Interventions: Biological: Vaccine: 2.6±0.8 x 10^10 vp/mL, 3 doses
- Cohort 4 (Experimental): Received three oral doses of 2.6±0.8 x 10^11 vp/mL Shigella flexneri 2a whole cell killed vaccine (Sf2aWC)
  Interventions: Biological: Vaccine: 2.6±0.8 x 10^11 vp/mL, 3 doses
- Placebo (Placebo Comparator): Received oral dose of placebo concurrent with Cohort 1 (one dose), 2, 3, or 4 (3 doses).
  Interventions: Biological: Placebo: 1-3 doses

INTERVENTIONS:
Biological: Vaccine: 2.6±0.8 x 10^8 vp/mL, 1 dose — Shigella flexneri 2a whole cell killed vaccine (Sf2aWC): 2.6±0.8 x 10^8 vp/mL administered on Day 0
  Arms: Cohort 1
Biological: Vaccine: 2.6±0.8 x 10^9 vp/mL, 3 doses — Shigella flexneri 2a whole cell killed vaccine (Sf2aWC): 2.6±0.8 x 10^9 vp/mL administered on Days 0, 28, and 56
  Arms: Cohort 2
Biological: Vaccine: 2.6±0.8 x 10^10 vp/mL, 3 doses — Shigella flexneri 2a whole cell killed vaccine (Sf2aWC): 2.6±0.8 x 10^10 vp/mL administered on Days 0, 28, and 56
  Arms: Cohort 3
Biological: Vaccine: 2.6±0.8 x 10^11 vp/mL, 3 doses — Shigella flexneri 2a whole cell killed vaccine (Sf2aWC): 2.6±0.8 x 10^11 vp/mL administered on Days 0, 28, and 56
  Arms: Cohort 4
Biological: Placebo: 1-3 doses — Placebo administered on Day 0 (if 1 dose) or Day 0, 28, and 56 (3 doses)
  Arms: Placebo

SUMMARY:
This is a research study about an experimental (investigational) oral inactivated whole cell Shigella flexneri 2a killed vaccine (Sf2aWC). Sf2aWC is a killed vaccine that is being made to prevent disease from Shigella., which causes bloody, watery diarrhea. Infants and children living in developing countries experience the greatest consequences of this disease. The purpose of this study is to find a dose of the vaccine that is safe, tolerable, and develops an immune response. About 82 healthy adults, ages 18-45, will participate in this study. This study will require volunteers to stay in the research facility for several nights for the first dose. Participants in Cohorts 2, 3, and 4 will not be required to stay overnight for the second and third doses. Participants will be assigned to receive 1 of 4 vaccine doses by mouth. Study procedures include: stool samples, blood samples and documenting side effects. Participants will be involved in study related procedures for about 8 months.

DETAILED DESCRIPTION:
Despite the public health burden of Shigella spp. on travelers, deployed soldiers and, most significantly, young children in the developing world, there is no licensed vaccine against Shigella. The rationale for using Shigella flexneri 2a whole cell killed vaccine (Sf2aWC), is that it is expected to be especially well tolerated by subjects. If Sf2aWC is safe and immunogenic, it may be combined with S. sonnei and S. flexneri 3a as the basis of a multivalent vaccine, because these three components should cover up to 80% of shigella infections in developing countries and over 90% in developed countries. This is a single site, Phase 1, double-blind, randomized, placebo-controlled, dose-escalation study in healthy adult subjects. Approximately 82 subjects will be enrolled into four separate cohorts and will be randomized to receive Sf2aWC or placebo. The placebo preparation will be bicarbonate buffer. Cohort 1 subjects will receive a single oral dose of Sf2aWC (2.6±0.8 x 10^8 vp/mL) or placebo. Dosing and 72 hours of supervised post-vaccination safety follow-up will be conducted in the Center for Immunization Research, Johns Hopkins School of Public Health (CIR) Inpatient Unit. Before enrolling subjects in subsequent cohorts, safety data from the previous Cohort(s) through Study Day 7 will be evaluated and reviewed by the Safety Review Committee (SRC). Cohorts 2, 3, and 4 participants will receive three doses of Sf2aWC vaccine or placebo at 0, 1 and 2 months. The first immunization will be administered in the CIR inpatient unit, followed by 72 hours of direct post-immunization observation. If after review by the SRC the first dose appears safe and well tolerated, subsequent doses will be administered on an outpatient basis. Safety will be assessed by solicited symptoms/subject memory aid and laboratory evaluations. Adverse events (AE)s will be graded according to standardized criteria. The immunogenicity outcome measures of interest include serum immunoglobulin G (IgG) and immunoglobulin A (IgA) antibodies by ELISA against S. flexneri 2a Lipopolysaccharide (LPS) and S. flexneri 2a invasive protein antigens (Ipa), cytokine assays, B and T cell memory responses, and vaccine-specific IgA responses. The proposed sample size of twenty per group in Cohorts 2, 3, and 4 would be sufficient to select the appropriate dose to move into the next study phase, providing that a difference in the immunogenicity between the two arms is 20% or greater. Participants will include 82 healthy adult male and female subjects, ages 18 to 45 inclusive. The primary objective of this study is to assess the safety and tolerability of Sf2aWC vaccine when administered in three oral doses over a range of dose levels in healthy adult subjects. The secondary objective is to assess the immunogenicity of the Sf2aWC vaccine over a range of doses in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, male or female, age 18 to 45 years (inclusive) at the time of enrollment.
* Completion and review of comprehension test (achieved >70% accuracy).
* Signed informed consent form.
* Available for the required follow-up period and scheduled clinic visits.
* Negative urine pregnancy test before each vaccination for female subjects of childbearing potential. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is also acceptable.

Exclusion Criteria:

* Presence of a significant medical or psychiatric condition that in the opinion of the investigator precludes participation in the study. Some medical conditions, that are adequately treated and stable, would not preclude entry into the study. These conditions might include stable asthma, hypertension or depression controlled with medication.
* Clinically significant abnormalities on physical examination.
* Clinically significant abnormalities in screening hematology, serum chemistry, or urinalysis as determined by PI or PI in consultation with Medical Monitor.
* History of febrile illness within 48 hours prior to vaccination.
* BMI <19 or >34.
* Positive blood test for HBsAG, hepatitis C virus (HCV), HIV-1, Human leukocyte antigen (HLA)-B27.
* Women currently nursing.
* History of reactive arthritis.
* Evidence of current excessive alcohol consumption
* Evidence of current drug use or drug dependence.
* Regular use of anti-diarrheal, anti-constipation, or antacid therapy (excluding use associated with spicy meals).
* Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis; loose or liquid stools on other than an occasional basis.
* Personal or family history of an inflammatory arthritis.
* History of allergy to soy products.
* History of microbiologically confirmed Shigella infection within 3 years.
* Prior receipt of experimental Shigella vaccine or live Shigella challenge within 3 years.
* Symptoms of travelers' diarrhea associated with travel to countries where Shigella or other enteric infections are endemic (most of the developing world) within 1 year prior to dosing.
* Occupation involving handling of Shigella bacteria currently, or in the past 3 years.
* History of diarrhea during the 7 days before vaccination.
* Use of antibiotics during the 7 days before vaccination.
* Use of proton pump inhibitors, H2 blockers, or antacids within 48 hours prior to dosing.
* Inability to comply with inpatient rules and regulations.
* Use of immunosuppressive and/or immunomodulative drugs such as corticosteroids or chemotherapeutics that may influence antibody development.
* Participation in research involving another investigational product (defined as receipt of investigational product or exposure to invasive investigational device) 30 days before planned date of first vaccination.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton D Harro, MD, ScM, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research (CIR) at Johns Hopkins School of Public Health (JHSPH), Baltimore, Maryland
  - Johns Hopkins University CIR Isolation Unit, Baltimore, Maryland

REFERENCES:
- [Result] Chakraborty S, Harro C, DeNearing B, Bream J, Bauers N, Dally L, Flores J, Van de Verg L, Sack DA, Walker R. Evaluation of the Safety, Tolerability, and Immunogenicity of an Oral, Inactivated Whole-Cell Shigella flexneri 2a Vaccine in Healthy Adult Subjects. Clin Vaccine Immunol. 2016 Apr 4;23(4):315-25. doi: 10.1128/CVI.00608-15. Print 2016 Apr. PMID 26865592

RESULTS

PARTICIPANT FLOW:
Period: Received Vaccination 1
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Placebo
Started | 5 | 20 | 20 | 20 | 17
Completed | 5 | 20 | 20 | 20 | 17
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Received Vaccination 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Placebo
Started | 5 | 20 | 20 | 20 | 17
Completed | 0 | 20 | 19 | 20 | 14
Not Completed | 5 | 0 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Illness | 0 | 0 | 0 | 0 | 1
Not completed — Not vaccinated per protocol | 5 | 0 | 0 | 0 | 2
Period: Received Vaccination 3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Placebo
Started | 0 | 20 | 19 | 20 | 14
Completed | 0 | 19 | 18 | 19 | 14
Not Completed | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject in Cohort 3 was randomized in error and did not receive the study product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Placebo | Total
Number analyzed (Participants) | 5 | 20 | 21 | 20 | 17 | 83
Age, Continuous [Mean (Full Range); unit: years] | 29 [25 to 34] | 31.7 [18 to 44] | 35.6 [18 to 45] | 32.3 [18 to 44] | 31.3 [20 to 45] | 32.6 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 3 | 8 | 5 | 24
  Male | 3 | 14 | 18 | 12 | 12 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 2 | 4
  Not Hispanic or Latino | 5 | 19 | 20 | 20 | 15 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 19 | 15 | 19 | 16 | 73
  White | 1 | 0 | 6 | 1 | 0 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Reactogenicity Per Subject and Treatment Group
Description: Local and systemic reactogenicity was assessed post-vaccination using targeted physical examinations, vital signs and clinical laboratory tests, and diary cards (completed following discharge daily through Day 7). Reactogenicity included: nausea, vomiting, fever, abdominal pain, abdominal cramping, bloating, malaise, headache, decreased appetite, generalized myalgias, chills, light-headedness, constipation, excessive flatulence, reactive arthritis, dysentery, loose stool, diarrhea, hypovolemia, joint pain, defecation urgency, and oral temperature.
Time Frame: 7 days after each vaccination (Day 0, Day 35, Day 63)
Population: Number may differ from overall number of participants analyzed if vaccination was not received.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 20 | 20 | 20
Participants
  After vaccination 1: None | 5 | 12 | 9 | 11
  After vaccination 1: Mild | 0 | 6 | 10 | 7
  After vaccination 1: Moderate | 0 | 0 | 1 | 2
  After vaccination 1: Severe | 0 | 2 | 0 | 0
  After vaccination 2: number analyzed (Participants) | 0 | 20 | 19 | 20
  After vaccination 2: None | 0 | 17 | 17 | 11
  After vaccination 2: Mild | 0 | 1 | 2 | 6
  After vaccination 2: Moderate | 0 | 2 | 0 | 3
  After vaccination 2: Severe | 0 | 0 | 0 | 0
  After vaccination 3: number analyzed (Participants) | 0 | 19 | 18 | 20
  After vaccination 3: None | 0 | 18 | 16 | 15
  After vaccination 3: Mild | 0 | 1 | 2 | 4
  After vaccination 3: Moderate | 0 | 0 | 0 | 1
  After vaccination 3: Severe | 0 | 0 | 0 | 0

2. Primary Outcome: Frequency of Unsolicited Adverse Events With a Reasonable Possibility That the Study Product Caused the Event
Time Frame: 6 months after final vaccination (Day 168 or Day 224)
Measure: Number; unit: adverse events
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Placebo
Number analyzed (Participants) | 5 | 20 | 20 | 20 | 17
adverse events
  Mild | 1 | 0 | 1 | 1 | 2
  Moderate | 0 | 0 | 0 | 1 | 1
  Severe | 0 | 0 | 0 | 0 | 0
  Total | 1 | 0 | 1 | 2 | 3

3. Secondary Outcome: Number and Percentage of Subjects in Cohort 3 With Positive Immunologic Response in Serum Lipopolysaccharide (LPS) Immunoglobulin A (IgA) Response From Baseline
Description: A positive immunological response is defined as an increase of 4-fold or more over the appropriate baseline value for ALS or an increase of more than 2-fold for serological responses (fold increases will be calculated to 1 decimal place). For all immunology variables, the raw values were first adjusted to the geometric mean of positive controls, and any values <0.15 were changed to 0.14. The fold-change in response was then calculated as the ratio of each value to the baseline value (so the minimum baseline value was 0.14). Specimens from vaccine recipients in Cohorts 1 and 2 were not tested for immunogenicity data and no data were collected.
Time Frame: 35 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3: Placebo: Received 3 oral doses of placebo for comparison with Cohort 3 subjects that received vaccine.
- Cohort 3: Vaccine: Received three oral doses of 2.6±0.8 x 10^10 vp/mL Shigella flexneri 2a whole cell killed vaccine (Sf2aWC)
  Vaccine: 2.6±0.8 x 10^10 vp/mL, 3 doses: Shigella flexneri 2a whole cell killed vaccine (Sf2aWC): 2.6±0.8 x 10^10 vp/mL administered on Days 0, 28, and 56
Arm/Group | Cohort 3: Placebo | Cohort 3: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 0 | 3
  Day 7: No | 5 | 17
  Pre-vaccination 2 (Day 28): number analyzed (Participants) | 5 | 19
  Pre-vaccination 2 (Day 28): Yes | 0 | 2
  Pre-vaccination 2 (Day 28): No | 5 | 17
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35: Yes | 0 | 2
  Day 35: No | 5 | 17

4. Secondary Outcome: Number and Percentage of Subjects in Cohort 4 With Positive Immunologic Response in Serum Lipopolysaccharide (LPS) Immunoglobulin A (IgA) Response From Baseline
Description: as for outcome 3
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 4: Placebo: Received 3 oral doses of placebo for comparison with Cohort 4 subjects that received vaccine.
- Cohort 4: Vaccine: Received three oral doses of 2.6±0.8 x 10^11 vp/mL Shigella flexneri 2a whole cell killed vaccine (Sf2aWC)
  Vaccine: 2.6±0.8 x 10^11 vp/mL, 3 doses: Shigella flexneri 2a whole cell killed vaccine (Sf2aWC): 2.6±0.8 x 10^11 vp/mL administered on Days 0, 28, and 56
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 0 | 13
  Day 7: No | 5 | 7
  Pre-vaccination 2 (Day 28): Yes | 0 | 3
  Pre-vaccination 2 (Day 28): No | 5 | 17
  Day 35: Yes | 0 | 9
  Day 35: No | 5 | 11
  Pre-vaccination 3 (Day 56): Yes | 1 | 4
  Pre-vaccination 3 (Day 56): No | 4 | 16
  Day 63: Yes | 0 | 10
  Day 63: No | 5 | 10

5. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Lipopolysaccharide (LPS) Immunoglobulin A (IgA) Response in Cohort 3
Description: S. flexneri 2a LPS were used as the ELISA antigens. Immunogenicity responses are presented for Cohorts 3 and 4 only. Specimens from vaccine recipients in Cohorts 1 and 2 were not tested for immunogenicity data and no data were collected. For all immunology variables, the raw values were first adjusted to the geometric mean of positive controls, and any values <0.15 were changed to 0.14.
Time Frame: 35 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 3: Placebo | Cohort 3: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 27 [20 to 36] | 23 [16 to 35]
  Day 7: number analyzed (Participants) | 5 | 19
  Day 7 | 31 [21 to 45] | 34 [22 to 55]
  Pre-vaccination 2 (Day 28): number analyzed (Participants) | 5 | 19
  Pre-vaccination 2 (Day 28) | 27 [18 to 41] | 28 [18 to 43]
  Day 35 | 26 [14 to 46] | 29 [19 to 47]

6. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Lipopolysaccharide (LPS) Immunoglobulin A (IgA) Response in Cohort 4
Description: as for outcome 5
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 240 [89 to 647] | 240 [89 to 647]
  Day 7 | 221 [62 to 784] | 757 [519 to 1105]
  Pre-vaccination 2 (Day 28) | 213 [79 to 576] | 345 [215 to 553]
  Day 35 | 281 [76 to 1038] | 560 [368 to 851]
  Pre-vaccination 3 (Day 56) | 278 [72 to 1065] | 376 [230 to 613]
  Day 63 | 252 [68 to 932] | 479 [315 to 727]

7. Secondary Outcome: Number and Percentage of Subjects in Cohort 3 With Positive Immunologic Response in Serum Lipopolysaccharide (LPS) Immunoglobulin G (IgG) Response From Baseline
Description: as for outcome 3
Time Frame: 16 weeks
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 0 | 0
  Day 7: No | 5 | 20
  Pre-vaccination 2 (Day 28): number analyzed (Participants) | 5 | 19
  Pre-vaccination 2 (Day 28): Yes | 1 | 3
  Pre-vaccination 2 (Day 28): No | 4 | 16
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35: Yes | 3 | 2
  Day 35: No | 2 | 17

8. Secondary Outcome: Number and Percentage of Subjects in Cohort 4 With Positive Immunologic Response in Serum Lipopolysaccharide (LPS) Immunoglobulin G (IgG) Response From Baseline
Description: as for outcome 3
Time Frame: 16 weeks
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 0 | 7
  Day 7: No | 5 | 13
  Pre-vaccination 2 (Day 28): Yes | 0 | 7
  Pre-vaccination 2 (Day 28): No | 5 | 13
  Day 35: Yes | 0 | 9
  Day 35: No | 5 | 11
  Pre-vaccination 3 (Day 56): number analyzed (Participants) | 5 | 19
  Pre-vaccination 3 (Day 56): Yes | 0 | 7
  Pre-vaccination 3 (Day 56): No | 5 | 12
  Day 63: Yes | 0 | 9
  Day 63: No | 5 | 11
  Week 16: Yes | 0 | 11
  Week 16: No | 5 | 9

9. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Lipopolysaccharide (LPS) Immunoglobulin G (IgG) Response in Cohort 3
Description: as for outcome 5
Time Frame: 35 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 3: Placebo | Cohort 3: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 1156 [255 to 5246] | 1388 [777 to 2482]
  Day 7 | 1388 [299 to 6450] | 1646 [955 to 2837]
  Pre-vaccination 2 (Day 28): number analyzed (Participants) | 5 | 19
  Pre-vaccination 2 (Day 28) | 1593 [365 to 6958] | 1464 [870 to 2464]
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35 | 1994 [391 to 10155] | 1790 [1056 to 3033]

10. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Lipopolysaccharide (LPS) Immunoglobulin G (IgG) Response in Cohort 4
Description: as for outcome 5
Time Frame: 16 weeks
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 2616 [763 to 8966] | 1530 [1013 to 2310]
  Day 7 | 2541 [757 to 8525] | 2571 [1777 to 3720]
  Pre-vaccination 2 (Day 28) | 2473 [848 to 7210] | 2514 [1770 to 3569]
  Day 35 | 2498 [847 to 7368] | 2997 [2099 to 4278]
  Pre-vaccination 3 (Day 56) | 2635 [781 to 8894] | 2884 [1971 to 4218]
  Day 63 | 2642 [801 to 8720] | 2969 [2070 to 4260]
  Week 16 | 2903 [814 to 10353] | 2722 [1771 to 4183]

11. Secondary Outcome: Number and Percentage of Subjects With Positive Immunologic Response in Serum Antibody From Lymphocytes Supernatant (ALS) Lipopolysaccharide (LPS) Immunoglobulin A (IgA) Response From Baseline
Description: as for outcome 3
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 4: Placebo | Cohort 3: Vaccine | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 5 | 20 | 20
Participants
  Day 7: Yes | 0 | 0 | 6 | 16
  Day 7: No | 5 | 5 | 14 | 4
  Pre-vaccination 2 (Day 28): number analyzed (Participants) | 5 | 5 | 19 | 20
  Pre-vaccination 2 (Day 28): Yes | 0 | 0 | 0 | 2
  Pre-vaccination 2 (Day 28): No | 5 | 5 | 19 | 18
  Day 35: number analyzed (Participants) | 5 | 5 | 19 | 20
  Day 35: Yes | 1 | 0 | 7 | 13
  Day 35: No | 4 | 5 | 12 | 7
  Pre-vaccination 3 (Day 56): number analyzed (Participants) | 5 | 5 | 18 | 19
  Pre-vaccination 3 (Day 56): Yes | 1 | 0 | 1 | 2
  Pre-vaccination 3 (Day 56): No | 4 | 5 | 17 | 17
  Day 63: number analyzed (Participants) | 4 | 5 | 18 | 20
  Day 63: Yes | 0 | 0 | 6 | 8
  Day 63: No | 4 | 5 | 12 | 12

12. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Antibody From Lymphocytes Supernatant (ALS) Lipopolysaccharide (LPS) Immunoglobulin A (IgA) Response From Baseline
Description: as for outcome 5
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 3: Placebo | Cohort 4: Placebo | Cohort 3: Vaccine | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 5 | 20 | 20
titer
  Baseline | 0.21 [0.14 to 0.32] | 0.21 [0.07 to 0.68] | 0.19 [0.15 to 0.24] | 0.22 [0.17 to 0.29]
  Day 7 | 0.18 [0.13 to 0.26] | 0.19 [0.11 to 0.32] | 0.47 [0.26 to 0.86] | 5.3 [2.58 to 11]
  Pre-vaccination 2 (Day 28): number analyzed (Participants) | 5 | 5 | 19 | 20
  Pre-vaccination 2 (Day 28) | 0.19 [0.10 to 0.34] | 0.16 [0.13 to 0.21] | 0.17 [0.14 to 0.19] | 0.27 [0.17 to 0.44]
  Day 35: number analyzed (Participants) | 5 | 5 | 19 | 20
  Day 35 | 0.22 [0.06 to 0.74] | 0.14 [0.14 to 0.14] | 0.58 [0.30 to 1.13] | 1.34 [0.73 to 2.47]
  Pre-vaccination 3 (Day 56): number analyzed (Participants) | 5 | 5 | 18 | 19
  Pre-vaccination 3 (Day 56) | 0.38 [0.06 to 2.29] | 0.14 [0.14 to 0.14] | 0.19 [0.13 to 0.28] | 0.25 [0.16 to 0.38]
  Day 63: number analyzed (Participants) | 4 | 5 | 18 | 20
  Day 63 | 0.31 [0.07 to 1.31] | 0.14 [0.13 to 0.15] | 0.42 [0.21 to 0.82] | 0.64 [0.35 to 1.17]

13. Secondary Outcome: Number and Percentage of Subjects With Positive Immunologic Response in Serum Antibody From Lymphocytes Supernatant (ALS) Lipopolysaccharide (LPS) Immunoglobulin G (IgG) Response From Baseline
Description: as for outcome 3
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 0 | 13
  Day 7: No | 5 | 7
  Pre-vaccination 2 (Day 28): Yes | 0 | 0
  Pre-vaccination 2 (Day 28): No | 5 | 20
  Day 35: Yes | 0 | 7
  Day 35: No | 5 | 13
  Pre-vaccination 3 (Day 56): number analyzed (Participants) | 5 | 19
  Pre-vaccination 3 (Day 56): Yes | 0 | 1
  Pre-vaccination 3 (Day 56): No | 5 | 18
  Day 63: Yes | 0 | 2
  Day 63: No | 5 | 18

14. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Antibody From Lymphocytes Supernatant (ALS) Lipopolysaccharide (LPS) Immunoglobulin G (IgG) Response
Description: as for outcome 5
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 0.65 [0.43 to 0.98] | 0.63 [0.41 to 0.96]
  Day 7 | 0.51 [0.24 to 1.09] | 4.93 [2.68 to 9.06]
  Pre-vaccination 2 (Day 28) | 0.42 [0.27 to 0.66] | 0.55 [0.37 to 0.81]
  Day 35 | 0.38 [0.12 to 1.16] | 1.32 [0.77 to 2.24]
  Pre-vaccination 3 (Day 56): number analyzed (Participants) | 5 | 19
  Pre-vaccination 3 (Day 56) | 0.36 [0.17 to 0.75] | 0.60 [0.37 to 0.98]
  Day 63 | 0.51 [0.18 to 1.44] | 0.94 [0.57 to 1.54]

15. Secondary Outcome: Number and Percentage of Subjects With Positive Immunologic Response in Invasion Plasmid Antigens B (IpaB) Lymphocytes Supernatant (ALS) Immunoglobulin A (IgA) Response From Baseline
Description: as for outcome 3
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 0 | 1
  Day 7: No | 5 | 19
  Pre-vaccination 2 (Day 28): Yes | 0 | 1
  Pre-vaccination 2 (Day 28): No | 5 | 19
  Day 35: Yes | 0 | 2
  Day 35: No | 5 | 18
  Pre-vaccination 3 (Day 56): number analyzed (Participants) | 5 | 19
  Pre-vaccination 3 (Day 56): Yes | 0 | 1
  Pre-vaccination 3 (Day 56): No | 5 | 18
  Day 63: Yes | 0 | 1
  Day 63: No | 5 | 19

16. Secondary Outcome: Geometric Mean Titer (GMT) of Invasion Plasmid Antigens B (IpaB) Lymphocytes Supernatant (ALS) Immunoglobulin A (IgA) Response
Description: Whole blood samples were collected for determination of ALS (antibody from lymphocytes supernatant). Immunogenicity responses are presented for Cohorts 3 and 4 only. Specimens from vaccine recipients in Cohorts 1 and 2 were not tested for immunogenicity data and no data were collected. For all immunology variables, the raw values were first adjusted to the geometric mean of positive controls, and any values <0.15 were changed to 0.14.
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 0.15 [0.13 to 0.17] | 0.20 [0.14 to 0.27]
  Day 7 | 0.15 [0.12 to 0.18] | 0.23 [0.17 to 0.32]
  Pre-vaccination 2 (Day 28) | 0.17 [0.12 to 0.24] | 0.20 [0.14 to 0.28]
  Day 35 | 0.14 [0.14 to 0.14] | 0.28 [0.16 to 0.48]
  Pre-vaccination 3 (Day 56): number analyzed (Participants) | 5 | 19
  Pre-vaccination 3 (Day 56) | 0.14 [0.14 to 0.14] | 0.19 [0.14 to 0.27]
  Day 63 | 0.14 [0.14 to 0.14] | 0.25 [0.15 to 0.42]

17. Secondary Outcome: Number and Percentage of Subjects With Positive Immunologic Response in Invasion Plasmid Antigen D (IpaD) Lymphocytes Supernatant (ALS) Immunoglobulin A (IgA) Response From Baseline
Description: as for outcome 3
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 0 | 1
  Day 7: No | 5 | 19
  Pre-vaccination 2 (Day 28): Yes | 0 | 0
  Pre-vaccination 2 (Day 28): No | 5 | 20
  Day 35: Yes | 0 | 2
  Day 35: No | 5 | 18
  Pre-vaccination 3 (Day 56): Yes | 0 | 1
  Pre-vaccination 3 (Day 56): No | 5 | 19
  Day 63: Yes | 0 | 0
  Day 63: No | 5 | 20

18. Secondary Outcome: Geometric Mean Titer (GMT) of Invasion Plasmid Antigen D (IpaD) Lymphocytes Supernatant (ALS) Immunoglobulin A (IgA) Response
Description: as for outcome 16
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | .14 [.14 to .14] | .17 [.14 to .21]
  Day 7 | .14 [.14 to .14] | .21 [.15 to .29]
  Pre-vaccination 2 (Day 28) | .15 [.13 to .17] | .18 [.14 to .23]
  Day 35 | .15 [.13 to .17] | .22 [.14 to .36]
  Pre-vaccination 3 (Day 56): number analyzed (Participants) | 5 | 19
  Pre-vaccination 3 (Day 56) | .14 [.14 to .14] | .19 [.14 to .27]
  Day 63 | .15 [.12 to .18] | .17 [.13 to .21]

19. Secondary Outcome: Number and Percentage of Subjects in Cohort 3 With Positive Immunologic Response in Fecal Immunoglobulin A (IgA) Response From Baseline
Description: as for outcome 3
Time Frame: 16 weeks
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 0 | 3
  Day 7: No | 5 | 17
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35: Yes | 0 | 3
  Day 35: No | 5 | 16
  Day 63: number analyzed (Participants) | 4 | 18
  Day 63: Yes | 1 | 4
  Day 63: No | 3 | 14
  Week 16: number analyzed (Participants) | 4 | 17
  Week 16: Yes | 0 | 4
  Week 16: No | 4 | 13

20. Secondary Outcome: Geometric Mean Titer (GMT) of Fecal Immunoglobulin A (IgA) Response in Cohort 3
Description: Immunogenicity responses are presented for Cohorts 3 and 4 only. Specimens from vaccine recipients in Cohorts 1 and 2 were not tested for immunogenicity data and no data were collected. For all immunology variables, the raw values were first adjusted to the geometric mean of positive controls, and any values <0.15 were changed to 0.14.
Time Frame: 16 weeks
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 3: Placebo | Cohort 3: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 21 [1.63 to 258] | 0.88 [0.39 to 1.94]
  Day 7 | 3.17 [0.22 to 45] | 1.02 [0.53 to 2.00]
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35 | 3.66 [0.30 to 45] | 0.68 [0.32 to 1.45]
  Day 63: number analyzed (Participants) | 4 | 18
  Day 63 | 5.64 [0.35 to 90] | 0.94 [0.32 to 2.71]
  Week 16: number analyzed (Participants) | 4 | 17
  Week 16 | 6.75 [0.48 to 94] | 1.74 [0.59 to 5.11]

21. Secondary Outcome: Number and Percentage of Subjects in Cohort 3 With Positive Immunologic Response in Total Immunoglobulin A (IgA) Response From Baseline
Description: as for outcome 3
Time Frame: 16 weeks
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 1 | 4
  Day 7: No | 4 | 16
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35: Yes | 0 | 1
  Day 35: No | 5 | 18
  Day 63: number analyzed (Participants) | 4 | 18
  Day 63: Yes | 1 | 5
  Day 63: No | 3 | 13
  Week 16: number analyzed (Participants) | 4 | 17
  Week 16: Yes | 0 | 5
  Week 16: No | 4 | 12

22. Secondary Outcome: Geometric Mean Titer (GMT) of Total Immunoglobulin A (IgA) Response in Cohort 3
Description: as for outcome 16
Time Frame: 16 weeks
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 3: Placebo | Cohort 3: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 0.23 [0.05 to 1.03] | 0.17 [0.02 to 0.57]
  Day 7 | 0.11 [0.02 to 0.57] | 0.14 [0.07 to 0.30]
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35 | 0.08 [0.01 to 0.45] | 0.08 [0.04 to 0.15]
  Day 63: number analyzed (Participants) | 4 | 18
  Day 63 | 0.09 [0.01 to 0.69] | 0.12 [0.05 to 0.33]
  Week 16: number analyzed (Participants) | 4 | 17
  Week 16 | 0.16 [0.04 to 0.62] | 0.29 [0.13 to 0.67]

23. Secondary Outcome: Number and Percentage of Subjects in Cohort 4 With Positive Immunologic Response in Total Immunoglobulin A (IgA) Response From Baseline
Description: as for outcome 3
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 0 | 6
  Day 7: No | 5 | 14
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35: Yes | 0 | 5
  Day 35: No | 5 | 14
  Day 63: number analyzed (Participants) | 5 | 18
  Day 63: Yes | 1 | 5
  Day 63: No | 4 | 13

24. Secondary Outcome: Geometric Mean Titer (GMT) of Total Immunoglobulin A (IgA) Response in Cohort 4
Description: as for outcome 16
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 0.63 [0.14 to 2.73] | 0.52 [0.32 to 0.85]
  Day 7 | 0.81 [0.17 to 3.74] | 1.31 [0.67 to 2.56]
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35 | 0.98 [0.14 to 6.69] | 0.87 [0.52 to 1.47]
  Day 63: number analyzed (Participants) | 5 | 18
  Day 63 | 0.66 [0.21 to 2.07] | 1.27 [0.59 to 2.70]

25. Secondary Outcome: Number and Percentage of Subjects in Cohort 4 With Positive Immunologic Response in Fecal Immunoglobulin A (IgA) Response From Baseline
Description: as for outcome 3
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
Participants
  Day 7: Yes | 2 | 7
  Day 7: No | 3 | 13
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35: Yes | 3 | 7
  Day 35: No | 2 | 12
  Day 63: number analyzed (Participants) | 5 | 18
  Day 63: Yes | 2 | 8
  Day 63: No | 3 | 10

26. Secondary Outcome: Geometric Mean Titer (GMT) of Fecal Immunoglobulin A (IgA) Response in Cohort 4
Description: as for outcome 20
Time Frame: 63 days
Population: Results were included for subjects that received each vaccination and with usable samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 4: Placebo | Cohort 4: Vaccine
Number analyzed (Participants) | 5 | 20
titer
  Baseline | 1.35 [0.25 to 7.39] | 2.11 [0.81 to 5.50]
  Day 7 | 2.06 [0.21 to 20] | 4.34 [1.18 to 16]
  Day 35: number analyzed (Participants) | 5 | 19
  Day 35 | 5.39 [0.47 to 61] | 4.01 [1.49 to 11]
  Day 63: number analyzed (Participants) | 5 | 18
  Day 63 | 3.98 [0.68 to 23] | 3.88 [0.97 to 15]

ADVERSE EVENTS:
Time Frame: 6 months after final vaccination (Day 168 for Cohort 1, or Day 224 for Cohort 2, 3, and 4)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/20 | 0/20 | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/20 | 0/20 | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/5 | 8/20 | 15/20 | 13/20 | 11/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=20) | Cohort 3 (N=20) | Cohort 4 (N=20) | Placebo (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Muscle strain (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 0 | 3
Blood urine present (Investigations) | 0 | 1 | 0 | 1 | 0
Eosinophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 3 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 2
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 3 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Vaginal infection (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No